CLINICAL TRIAL: NCT02414113
Title: A Blinded, Prospective Non-Interventional Observational Study for the Evaluation of a GVHD Negative Outcome Score (GNOS) in Matched Unrelated or Haploidentical Hematopoietic Stem Cell Transplant
Brief Title: Study for the Evaluation of a GVHD Negative Outcome Score (GNOS) in Matched Unrelated or Haploidentical Hematopoietic Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Predictive BioDiagnostics, LLC (Unknown); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: 201312100
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hematopoietic Stem Cell Transplantation; Stem Cell Transplantation, Hematopoietic; Transplantation, Hematopoietic Stem Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — -At the time of HLA confirmatory typing, 24 mL of whole blood will be collected from all potential donors who agree to participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low GNOS donors
- High GNOS donors

SUMMARY:
Before considering high-GVHD Negative Outcome Score (GNOS) donor selection for routine clinical practice, this blinded prospective study will be carried out for assessment of severe GVHD (graft-versus-host-disease) reduction associated with selecting high-GNOS donors for allogeneic hematopoietic peripheral blood stem cell transplant. The objective of this prospective study is to show: (a) that GVHD reductions and donor availabilities as observed in the retrospective studies also apply to prospective samples that are collected and processed from on-going matched unrelated transplants, and (b) that high-GNOS donor selection readily fits into today's donor selection process, such as to facilitate access to the benefits of GVHD reduction. The prospective study is designed to be blinded, and will not involve specific donor selection nor any influence on clinical management or decision making by application of the GNOS technology.

To determine if some GNOS models perform better than others across different clinical centers, or across different recipient / donor attributes, 4 different specific GNOS models will be evaluated. Bootstrap computational analyses have been carried out on the retrospective data for the 4 GNOS models and will be tested and validated in this prospective study.

DETAILED DESCRIPTION:
Enrollment of the recipient will occur prior to the unrelated donor search or haploidentical donor identification.

FOR UNRELATED DONORS:

When the unrelated donor search is formalized, the study team will submit a study participation request document to the NMDP for all potential donors that are being evaluated for an enrolled recipient. These documents will be relayed to the appropriate donor centers by the NMDP. This document informs the donor center that the potential donor's participation in this trial is being requested. The donor center then will approach the potential donor about participation in the trial. If the potential donor consents to participate, the required donor study samples will be obtained and shipped to the appropriate labs. This will conclude the potential donor's physical participation in the trial. The donor consent will be kept at the donor center and will not be provided to the investigator.

FOR HAPLOIDENTICAL DONORS:

Haploidentical donors will be identified by the transplant team caring for the recipient, and will follow the site's standard procedures for identification, HLA typing, and medical clearance for stem cell donation. Haploidentical donors will be approached by the transplant team or the study coordinator about participation in the trial. If the potential donor consents to participate, the required donor study samples will be obtained and shipped to the appropriate lab for processing prior to the start of growth factor for stem cell mobilization or prior to stem cell collection via bone marrow harvest.

FOR ALL DONORS:

At the time of HLA confirmatory typing, 24 mL of whole blood will be collected from donors.

ELIGIBILITY:
Eligibility Criteria Prior to Unrelated Donor Search / Haploidentical Donor Identification:

* Recipient must be between 18 and 70 years of age, inclusive
* Recipient must be undergoing unrelated or haploidentical stem cell donor search with one or more potential donors being requested for confirmatory typing and study samples.
* Recipient must be able to understand and willing to sign written informed consent document

Eligibility Criteria on Day 0:

* Selected donor must have agreed to participate in the trial and samples for GNOS must have been received and processed.
* If MUD donor, selected donor must not be a C-antigen mismatch with the recipient (C-allele mismatch donor-recipient pairs are eligible).
* Recipient must not have received alemtuzumab as part of stem cell conditioning regimen.
* Recipient must not undergo transplantation with ex vivo T-cell depleted stem cells.
* If MUD donor, recipient must receive a myeloblative stem cell conditioning (MAC) regimen per CIBMTR (Center for International Blood and Marrow Transplant Research) criteria. Patients that receive only low intensity, non-myeloablative conditioning regimen will be excluded.
* If haploidentical donor, recipient must receive standard MAC or RIC-conditioning with post-transplant Cytoxan GVHD prophylaxis given on Days +3 and +4.

Enrollment will occur prior to the unrelated donor search. Following donor selection, if the recipient does not meet the eligibility criteria listed for Day 0 or if the recipient does not proceed to stem cell transplantation within 12 months of enrollment, the donor/recipient pair will be non-evaluable for the study objectives. Non-evaluable donor/recipient pairs will be removed from trial and replaced.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Matched unrelated hematopoietic stem cell transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Rates of grade III-IV aGVHD (acute graft-versus-host disease) in hematopoietic stem cell transplantation (HSCT) performed with high GNOS versus low GNOS donors | 100 days after HSCT
  * "GNOS" refers to PBD's proprietary "GVHD Negative Outcome Score" technology for reduction of grades III & IV aGVHD through donor selection. GNOS is a gene expression-based signature of lower donor allo-reactivity such that transplanted cells from donors displaying higher GNOS will exhibit less allo-reactivity against recipient tissues, therefore decreasing the incidence of severe GVHD. GNOS is determined from pre-transplant, pre-mobilization gene expression profiling of donor CD4 cells from a blood draw.
  * Incidence and severity of acute GVHD will be assessed based on the modified Glucksberg criteria and Seattle criteria. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s) as per standard of care.

SECONDARY OUTCOMES:
Overall survival in HSCT performed with high GNOS versus low GNOS donor who experienced Grades 0-II and Grades III-IV aGVHD during the first 100 days after HSCT | 3 months
  -Overall survival (OS) is defined as the date of transplant to the date of death from any cause.
Performance of 4 pre-defined GNOS models | 100 days after HSCT
  * The main variables' association of interest, for any of the 4 outcome predictive models being employed, is recipient aGVHD Grades {0, I, II} exclusive-or Grades {III-IV} vs. donor GNOS level. The analyses will be done separately for each of the 4 different outcome predictive models that have been employed in the study.
  * The GNOS values from each of 4 models will be determined by PBD and will be kept confidential and blinded from the investigators. PBD will not know the recipient health data (GVHD occurrence, PFS, OS, etc.) when the GNOs analysis is performed. Thus, a given donor's GNOS values from the 4 different models and the corresponding recipient's outcomes will not be correlated until after unblinding.
Relapse rates after HSCTs performed with high GNOS versus low GNOS donors | 1 year
  -A patient will be considered relapsed when there is a recurrence of the original malignant disease after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - UNC Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu